CLINICAL TRIAL: NCT01344161
Title: Effect of Vitamin D on Metabolic Profile in Overweight or Obese Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRCT138809092709N2
Record Dates: First submitted 2011-04-18; First posted 2011-04-28 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Overweight; Obesity
Keywords: Vitamin D; Metabolic profile; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Lactose; Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactose (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Vitamin D (Experimental)
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: Placebo — dosage form:lactose dosage: 25 micrograms frequency: every day duration: 12weeks
  Other Names: Lactose
  Arms: Lactose
Dietary Supplement: vitamin D — dosage form:cholecalciferol dosage: 25 micrograms (1000 International Unit) frequency: every day duration: 12weeks
  Other Names: Cholecalciferol
  Arms: Vitamin D

SUMMARY:
The investigators investigated the effect of vitamin D3 supplementation on metabolic profile (anthropometric measures, blood pressure Lipids, lipoproteins and glycemic indices) in overweight or obese women.

DETAILED DESCRIPTION:
Vitamin D deficiency is a worldwide health problem and is determined as a risk factor in Cardiometabolic disorders including Cardiovascular disease, Metabolic syndrome, and type 2 diabetes mellitus. The investigators investigated the effect of vitamin D3 supplementation on metabolic profile in overweight or obese women.

A double blind randomized clinical trial was conducted in 77 premenopause overweight or obese women. Participants were classified into two groups : vitamin D supplementation [1000 IU/day as cholecalciferol tablets (n=39)] or placebo (n=38). Vein blood samples were taken after at least 12 hours overnight fasting. Selected anthropometric measures, blood pressure Lipids, lipoproteins and glycemic indices were measured at baseline and after 12 weeks. Body fat mass was determined using BIA. Also the investigators assessed dietary intake using 24 hours food recall and semi-quantitative food frequency and physical activity using IPAQ questionnaires.

The investigators conducted the study between October 2009 and March 2010 at the Medical school, Tehran, Iran. Recruitment began in October 2009 via advertisements and was terminated in October 2009. The investigators excluded patients with a history of Cardiovascular disease, Liver disease, Gastrointestinal disease, Kidney disease, diabetes mellitus, and Osteoporosis. Moreover, pregnancy, lactation, vegetarianism, and intake of dietary supplements were the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-50 years old
* Premenopause
* BMI ≥25

Exclusion Criteria:

* Cardiovascular disease
* Liver disease
* Gastrointestinal disease
* Kidney disease
* Diabetes mellitus
* Osteoporosis
* Pregnancy
* Lactation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farzad Shidfar, PhD, Study Director — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Salehpour A, Shidfar F, Hosseinpanah F, Vafa M, Razaghi M, Amiri F. Does vitamin D3 supplementation improve glucose homeostasis in overweight or obese women? A double-blind, randomized, placebo-controlled clinical trial. Diabet Med. 2013 Dec;30(12):1477-81. doi: 10.1111/dme.12273. Epub 2013 Jul 27. PMID 23822797
- [Derived] Salehpour A, Hosseinpanah F, Shidfar F, Vafa M, Razaghi M, Dehghani S, Hoshiarrad A, Gohari M. A 12-week double-blind randomized clinical trial of vitamin D(3) supplementation on body fat mass in healthy overweight and obese women. Nutr J. 2012 Sep 22;11:78. doi: 10.1186/1475-2891-11-78. PMID 22998754

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In November 2009 we distributed advertisements in campus of Tehran University of Medical Sciences (TUMS) and invited all female students and employee to participate in our study.
Groups:
- Lactose: In placebo group women used a pill of 25 microgram lactose every day for 12-weeks.
- Vitamin D: In vitamin D group women used a pill of 25 microgram cholecalciferol every day for 12-weeks.
Period: Overall Study
Arm/Group | Lactose | Vitamin D
Started | 43 | 42
Completed | 38 | 39
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactose | Vitamin D | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 39 | 77
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.9 (7) | 37 (8) | 38 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 38 | 39 | 77

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Fat Mass
Description: Body composition was assessed by Bioelectrical Impedance Analysis (model 4000; Body Stat Quad Scan, Douglas Isle of Man, British Isles).The principle of measuring the flow of current through the body is dependent on the frequency applied. At low frequencies, the current cannot bridge the cellular membrane and will pass predominantly through the extra-cellular space. At higher frequencies penetration of the cell membrane occurs and the current is conducted by both the extra-cellular water (ECW) and intra-cellular water (ICW).FFM can be estimated because FFM is primarily composed of water.
Time Frame: 3 months minus baseline
Population: We assessed body composition by Bioelectrical Impedance Analysis (model 4000; Body Stat Quad Scan, Douglas Isle of Man, British Isles).
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Vitamin D: 25 microgram cholecalciferol
- Placebo: 25 microgram lactose
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 39 | 38
kg | -2.7 (2) | -0.4 (2)
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; An analysis of covariance (ANCOVA) was used to adjust mean differences on all variables; Mean Difference (Net) = 0.05

2. Primary Outcome: Change in Glucose Concentrations
Time Frame: 3 months minus baseline
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 39 | 38
mmol/L | -0.28 (0.4) | -0.65 (.4)

3. Primary Outcome: Change in Post Load Glucose Concentrations
Description: It was performed 2 hours after 75g oral glucose tolerance test (75-OGTT).
Time Frame: 3 months minus baseline
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 39 | 38
mmol/L | -0.29 (0.9) | -0.3 (1.1)

4. Primary Outcome: Change in Insulin Concentrations
Time Frame: 3 months minus baseline
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 39 | 38
pmol/L | -24.8 (20.2) | -19 (23.3)

ADVERSE EVENTS:
Arm/Group | Lactose | Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 0/38 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No